CLINICAL TRIAL: NCT02074085
Title: Measuring the Incidence of Hospital Readmissions, Caused by Adverse Drug Events (ADE) Due to Anticoagulants in Vzw Jessa Hospital (Belgium)
Brief Title: Measuring the Incidence of Hospital Readmissions Based on Adverse Drug Events
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, prof. dr. Neree Claes, prof. dr., Hasselt University
Other Study IDs: 14.05/APO14.01
Record Dates: First submitted 2014-02-25; First posted 2014-02-28 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Incidence of Readmissions; ADE's Due to Anticoagulants

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
An ADE is defined as harm caused by a drug or the inappropriate use of a drug. Retrospective record reviews in several countries have shown that anticoagulants frequently lead to hospital readmissions. In this study a hospital readmission is defined as an admission to the emergency department of the Jessa hospital. The objective of this study is to determine the incidence of one week and 30-day readmissions caused by (preventable) ADE's due to anticoagulants.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who received an anticoagulant on their last day of admission
2. Patients who were readmitted within 30 days
3. Patients who were diagnosed using the pathology registration of the emergency department of the Jessa hospital

Exclusion Criteria:

1. Patients who didn't receive an anticoagulant on their last day of admission
2. Patients who were not readmitted within 30 days
3. Patients who were not diagnosed using the pathology registration of the emergency department of the Jessa hospital
4. Patients with missing data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who received an anticoagulant on their last day of admission
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
incidence of readmissions within one week caused by ADE's due to anticoagulants | up to one week
incidence of readmissions within 30 days caused by ADE's due to anticoagulants | up to 1 month
incidence of preventable ADE's leading to readmission | week 1, month 1

CONTACTS AND LOCATIONS:
Overall Officials: Martijn Droogmans, pharmacist, Study Chair — Jessa Hospital; Kristel Marquet, drs, Study Chair — Hasselt University; Janne Theuwissen, pharmacist, Study Chair — Jessa Hospital
Locations (1):
- Jessa Ziekenhuis, Hasselt, Belgium